CLINICAL TRIAL: NCT06192550
Title: Functional Usability and Feasibility Testing of the Profound Matrix™ System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Candela Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUFT2002
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-10

CONDITIONS: Wrinkle; Acne Scars - Mixed Atrophic and Hypertrophic
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Group 1: Matrix Pro (Experimental): Subjects undergoing treatment with the Matrix Pro applicator.
  Interventions: Device: Profound Matrix™ System
- Group 2: Sublime/Sublative (Experimental): Subjects undergoing treatment with either 1) Sublime applicator only, 2) Sublative RF applicator only, 3) Combined treatment of Sublime and Sublative RF applicators.
  Interventions: Device: Profound Matrix™ System
- Modified Matrix Pro (Experimental): Subjects undergoing treatment with a Matrix Pro Modified applicator with lower RF power settings.
  Interventions: Device: Profound Matrix™ System

INTERVENTIONS:
Device: Profound Matrix™ System — Study subjects will be treated with the Profound Matrix System

SUMMARY:
This is a non-randomized, multi-center, open-label clinical trial evaluating the efficacy and clinical feasibility of the Profound Matrix device for electrocoagulation and for treatment of wrinkles and acne scars. Subjects will receive up to three (3) treatments with the Matrix Pro applicator or up to five (5) treatments with the Sublime and/or Sublative Radiofrequency (RF) applicators.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male or Female
2. Age 18 to 75
3. Subjects seeking treatment for facial, abdominal, or back wrinkles reduction, skin texture improvement and/or acne scars appearance improvement and willing to undergo RF treatments for improvement
4. Presence of at least mild wrinkles or mild acne scars or uneven skin texture, as assessed by the Investigator
5. Willingness to provide signed, informed consent to participate in the study
6. Willingness to allow photography of treated areas, and to release their use for scientific/educational and/or promotional purposes

Exclusion Criteria:

1. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
2. Pacemaker or internal defibrillator or any active electrical implant anywhere in the body
3. Superficial metal or other implants in the treatment area, except superficial dental implants, unless these implants can be removed or covered with rolled gauze during treatment
4. Current skin cancers in the treatment area or history of melanoma
5. History of current cancer and subject has undergone chemotherapy within the last 12 months
6. Severe concurrent conditions, such as cardiac disorders
7. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
8. Herpes Simplex Virus (HSV) in the intended treatment area unless treated following a prophylactic regimen
9. Poorly controlled endocrine disorders such as diabetes
10. Active skin condition in the treatment area such as sores, psoriasis, eczema, or rash, open wounds, and severe active inflammatory acne.
11. History of abnormal wound healing, keloid, or hypertrophic scar formation, as well as very dry and fragile skin
12. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitis disorders
13. Known allergy to lidocaine, tetracaine, Xylocaine, epinephrine or ProNox (nitrous oxide (laughing gas))
14. Patients on systemic corticosteroid therapy in past six months
15. Is taking medication(s) for which sunlight is a contraindication
16. Tattoos or permanent makeup in the intended treatment area
17. Excessively tanned skin
18. Subjects with pigmented lesions that are considered not acceptable by the study investigator or any condition that, in the investigator's opinion, would make it unsafe to treat.
19. Subject has hair and is unwilling to have hair removed from the treatment area
20. Subjects has undergone facelift in the last 12 months
21. Subject has undergone aesthetics treatments/procedures (e.g. facial resurfacing and deep chemical peeling) within the last 4 months) within the intended to treat area
22. Subject has undergone Botox in the treatment area within the last 3 months
23. Subject has non-permanent filler in the last 3 months within the intended to treat area
24. Subject has permanent filler (e.g. silicone) within the intended to treat area
25. Subject has absorbable facial threads within the last 2 years within the intended to treat area
26. Subject has non-absorbable facial threads within the intended to treat area aa. Subject is using a topical in the treatment area that the Investigator's deems the subject unsuitable for the study.

bb. In the opinion of the Investigator, the subject is unwilling or unable to adhere to the study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Investigator Global Aesthetic Improvement Scale (GAIS): Perceived Improvement in Overall Appearance | 3 months post final treatment
  Perceived improvement in overall appearance according to the 5-point Global Aesthetic Improvement Scale from -1= Worse to 3= Very Much Improved as assessed by investigator at study endpoint

SECONDARY OUTCOMES:
Subject Global Aesthetic Improvement Scale (GAIS): Perceived Improvement in Overall Appearance | 3 months post final treatment
  Perceived improvement in overall appearance according to the 5-point Global Aesthetic Improvement Scale from -1= Worse to 3= Very Much Improved as assessed by subject at study endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Konika Schallen, MD, Principal Investigator — Candela Medical
Locations (5):
- United States (4):
  - Candela Institue for Excellence, Marlborough, Massachusetts
  - NY Derm, New York, New York
  - OptiSkin, New York, New York
  - Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
- Syneron Medical, Yokneam Illit, Israel

IPD SHARING:
Plan to Share IPD: No